CLINICAL TRIAL: NCT02911259
Title: Suction on Post-Operative Chest Tubes After Video-Assisted Thoracoscopic Surgery Lobectomy for Presumed or Confirmed Primary Lung Cancer - At Which Level?
Brief Title: Suction on Post-Operative Chest Tubes
Acronym: SPOCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Medela AG (Industry)
Responsible Party: Principal Investigator, Bo Laksáfoss Holbek, Medical doctor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-15008900
Record Dates: First submitted 2016-02-23; First posted 2016-09-22 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Post-operative suction is set to -2 cmH2O.
  Interventions: Device: Suction is set to -2 cmH2O
- Group 2 (Active Comparator): Post-operative suction is set to -10 cmH2O (standard treatment).
  Interventions: Device: Suction is set to -10 cmH2O

INTERVENTIONS:
Device: Suction is set to -2 cmH2O — Post-operative suction is set to -2 cmH2O (intervention).
  Arms: Group 1
Device: Suction is set to -10 cmH2O — Post-operative suction is set to -10 cmH2O (standard treatment).
  Arms: Group 2

SUMMARY:
The level of suction on post-operative chest tubes after video-assisted thoracoscopic surgery (VATS) lobectomy for lung cancer has previously shown to affect duration of drainage. These results, however, are based on traditional drainage systems with water seal and need to be confirmed using digital drainage systems.

Hypothesis: Suction of -2 cmH2O is equal to or superior compared with standard suction of -10 cmH2O when looking at chest tube duration and complications.

ELIGIBILITY:
Inclusion Criteria:

* Speaks and understands Danish.
* Referred for planned VATS lobectomy for confirmed or suspected primary lung cancer.

Exclusion Criteria:

* Cannot cooperate or unable to give consent.
* Chronic drain carrier.
* Planned open procedure.
* Planned resection of additional wedge, additional lobe or thoracic wall.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-14 (Actual)

PRIMARY OUTCOMES:
Chest tube duration through study completion, an average of 3 days. | Through study completion, an average of 3 days.
  Time from intraoperative chest tube placement to it's removal.

SECONDARY OUTCOMES:
Time to removal criteria have been fulfilled up to 24 hours | Duration from the post-operative chest tube has been placed, until it's potential removal.
  Chest tubes can be removed when the patient has been mobilized and the air leakage has not superceeded 20 mL/min in 12 hours and fluid production has not superceded 500 mL in 24 hours.
Number of participants with prolonged air leak | Through study completion, an average of 7 days
Number of participants requiring treatment for prolonged air leak. | Through study completion, an average of 14 days
Number of participants requiring treatment for subcutaneous emphysema. | Through study completion, an average of 14 days
Number of participants with pneumonia or empyema. | Through study completion, an average of 21 days
Length of stay. | Through study completion, an average of 3 days
Number of participants with other respiratory problems. | Through study completion, an average of 30 days
Number of participants requiring readmission for thoracic surgical complications. | Through study completion, an average of 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Bo L. Holbek, MD, Principal Investigator — Rigshospitalet, Denmark; Merete Christensen, MD, Study Director — Rigshospitalet, Denmark; Jesper Ravn, MD, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marshall MB, Deeb ME, Bleier JI, Kucharczuk JC, Friedberg JS, Kaiser LR, Shrager JB. Suction vs water seal after pulmonary resection: a randomized prospective study. Chest. 2002 Mar;121(3):831-5. doi: 10.1378/chest.121.3.831. PMID 11888968
- [Background] Cerfolio RJ, Bryant AS. The management of chest tubes after pulmonary resection. Thorac Surg Clin. 2010 Aug;20(3):399-405. doi: 10.1016/j.thorsurg.2010.04.001. PMID 20619231
- [Background] Brunelli A, Beretta E, Cassivi SD, Cerfolio RJ, Detterbeck F, Kiefer T, Miserocchi G, Shrager J, Singhal S, Van Raemdonck D, Varela G. Consensus definitions to promote an evidence-based approach to management of the pleural space. A collaborative proposal by ESTS, AATS, STS, and GTSC. Eur J Cardiothorac Surg. 2011 Aug;40(2):291-7. doi: 10.1016/j.ejcts.2011.05.020. PMID 21757129
- [Background] Gottgens KW, Siebenga J, Belgers EH, van Huijstee PJ, Bollen EC. Early removal of the chest tube after complete video-assisted thoracoscopic lobectomies. Eur J Cardiothorac Surg. 2011 Apr;39(4):575-8. doi: 10.1016/j.ejcts.2010.08.002. Epub 2010 Sep 15. PMID 20833554
- [Background] Cerfolio RJ, Varela G, Brunelli A. Digital and smart chest drainage systems to monitor air leaks: the birth of a new era? Thorac Surg Clin. 2010 Aug;20(3):413-20. doi: 10.1016/j.thorsurg.2010.03.007. PMID 20619233
- [Background] Pompili C, Detterbeck F, Papagiannopoulos K, Sihoe A, Vachlas K, Maxfield MW, Lim HC, Brunelli A. Multicenter international randomized comparison of objective and subjective outcomes between electronic and traditional chest drainage systems. Ann Thorac Surg. 2014 Aug;98(2):490-6; discussion 496-7. doi: 10.1016/j.athoracsur.2014.03.043. Epub 2014 Jun 4. PMID 24906602
- [Derived] Holbek BL, Christensen M, Hansen HJ, Kehlet H, Petersen RH. The effects of low suction on digital drainage devices after lobectomy using video-assisted thoracoscopic surgery: a randomized controlled trialdagger. Eur J Cardiothorac Surg. 2019 Apr 1;55(4):673-681. doi: 10.1093/ejcts/ezy361. PMID 30445572